CLINICAL TRIAL: NCT01068691
Title: Blood Pressure Control and Arterial Properties After Surgical Treatment of Type A Thoracic Aortic Dissection or Haematoma
Brief Title: Arterial Properties of Thoracic Aorta Disease
Acronym: ao_diss
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Pr Jean-Philippe BAGUET, Laboratoire Hypertension Artérielle-Pôle cardiovasculaire et thoracique
Other Study IDs: 706; 2007-A01422-51 (Registry Identifier: AFSSAPS)
Record Dates: First submitted 2009-06-22; First posted 2010-02-15 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Blood Pressure
Keywords: aortic dissection; ambulatory blood pressure; obstructive sleep apnea syndrome; patients undergoing surgery for a dissection of the thoracic aorta
MeSH Terms: conditions — Aortic Dissection; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples for inflammation, oxidative stress and collagen markers
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Ambulatory blood pressure monitoring (to evaluate the level of blood pressure) — * Ambulatory blood pressure monitoring (to evaluate the level of blood pressure)
  * Blood pressure
  * Obstructive sleep apnea syndrome (OSAS)
  * Carotid-to-femoral pulse wave velocity (PWV)
  * Biological parameters

SUMMARY:
A dissecting or intramural haematoma of the thoracic aorta (AH) is a haemorrhage that dissects the aortic wall. An entry point is detected at an intimal tear, ulcer or plaque rupture via imaging in almost 50% of cases. AH occurs in older patients than those with AD and develops on atheromatous lesions with parietal ulcers, most often in cases of poorly managed, pre-existing hypertension (HTN). Type A AHs, which affect the ascending aorta, frequently progress towards an AD with a high risk of mortality, and represent a surgical indication.

Patients who have presented AD or AH, whether they have been operated or not, must undergo prolonged monitoring. This involves both clinical and radiological checks to ensure that blood pressure is properly monitored, that the parietal lesions have receded and that there are no complications.

HTN is a recognized risk factor for the onset of AD and systolic blood pressure must be brought down to between 100 and 120 mmHg perioperatively. Furthermore, HTN is also a risk factor for the rupture of unoperated type B AD. Despite this, only two studies have looked at BP management in AD patients. The first, carried out among chronic type A or B AD patients revealed that closer monitoring of blood pressure levels at home led to a better long-term prognosis. Another study revealed a 60% prevalence of non-managed clinical HTN among 40 chronic AD patients.

Whilst frequent, regular aortic wall monitoring via imaging methods (CT or MRI) is recommended after thoracic AD surgery, there is no precise recommendation as to the method of BP monitoring in very high-risk patients. A BP level of 135/80 mmHg has been suggested as a maximum limit for patients having been operated for AD. In order to achieve this, antihypertensives of several therapeutic classes must be used, with beta-blockers as a priority. The same can be said for AH, as it has been demonstrated that the absence of beta-blocker treatment is a predictive factor for poor progress.

Increased aortic stiffness can cause increased systolic blood pressure and is recognized as an independent cardiovascular risk factor. This stiffness can be detected by measuring the carotid-to-femoral pulse wave velocity (PWV). No study has as yet focused on assessing aortic stiffness in patients who have undergone AD or AH surgery.

Obstructive sleep apnea syndrome (OSAS) in thoracic AD patients is highly prevalent, and respiratory events that occur are more severe. This has prompted some to suggest that systematic detection of OSAS after AD should be carried out. No findings have yet been published about patients who have undergone AH surgery.

DETAILED DESCRIPTION:
Main objective:

* To evaluate the level of blood pressure control using ambulatory blood pressure monitoring in patients who have undergone surgery for a type A thoracic AD or AH.

Secondary objectives:

* To study aortic stiffness within this patient population and determine its predictive parameters.
* To determine the prevalence of OSAS among this patient population and study the relationship between respiratory data and blood pressure values.
* To determine the respective roles of blood pressure level, aortic stiffness, and respiratory and biological parameters upon the postoperative aortic diameters of patients who have undergone surgery for type A thoracic AD or AH.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients aged 18 or over who:

* benefit from the French social security system
* will be monitored as outpatients
* have given their written consent to participate in this study
* have been operated over 6 months ago for a type A thoracic AD or AH at Grenoble University Hospital in the period from 1 January 1990 to 30 June 2007
* are able to travel to Grenoble University Hospital

Exclusion Criteria:

* Bedridden or reduced mobility patients.
* Patients whose physical or psychological condition could affect their informed consent and compliance with the requirements of the protocol.
* Adult patients protected by the law (article L1121-8 of the French Public Health Code).
* Individuals serving a prison sentence (article L1121-8 of the French Public Health Code).
* Women who are pregnant, have recently given birth or are breastfeeding.
* Patients in the terminal phase of a serious illness.
* Individuals serving a prison sentence as a result of a legal or administrative ruling, or individuals receiving legal protection.
* Children.
* Patients taking part in another study.
* Individual who is not part of the social security system or who does not benefit from it.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a pilot, descriptive and single-centre study.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Ambulatory blood pressure monitoring | the same day as inclusion

SECONDARY OUTCOMES:
Aortic stiffness, Aortic diameters | the same day as inclusion
polysomnography to research Sleep apnea | within 2 months

CONTACTS AND LOCATIONS:
Overall Officials: jean-philippe baguet, Pr, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, France